CLINICAL TRIAL: NCT04719611
Title: Detection of Probiotic Strains in Vaginal Swabs Collected From Healthy Adults Consuming a Probiotic Supplement: a Pilot Study (VSS)
Brief Title: Detection of Probiotic Strains in Vaginal Swabs Collected From Healthy Women
Acronym: VSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Collaborators: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: L-021
Record Dates: First submitted 2021-01-15; First posted 2021-01-22 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Probiotics; Strain recovery; Vaginal swab; Persistence
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: interventional, single-arm, open-label, pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy Women (Experimental): Healthy women between the ages of 18-40 years will be given a probiotic supplement to evaluate the detection and persistence of the strains in biological samples.
  Interventions: Dietary Supplement: Probiotic

INTERVENTIONS:
Dietary Supplement: Probiotic — Healthy women receive a probiotic supplement containing 6 x 10^9 colony-forming units/capsule of Bifidobacterium and Lactobacillus strains.

SUMMARY:
The aim of this trial is to detect the presence of various probiotic strains in vaginal swabs of healthy women orally consuming a probiotic supplement for 4 weeks.

DETAILED DESCRIPTION:
Participants recruited from the university community in the Southeast U.S. will participate in a pilot, open-label interventional study for approximately 6 weeks following obtainment of informed consent. Participants will be asked to maintain their usual diets with the exception of probiotic supplements, probiotic fortified products or foods with added fiber supplements.

On the first day of the study, participants will take part in a 1-week pre-baseline period where they will begin daily questionnaires inquiring about gastrointestinal symptoms, stool form and number, stress, and medications taken.

On the first day of the intervention period (Day 1), participants will self collect a baseline vaginal swab sample, a skin swab, a vaginal pH swab, and a stool sample. Participants will consume 2 capsules every morning and 2 capsules every evening for four weeks (from D1 to D28).

Participants will self collect a vaginal swab sample, a skin swab, a vaginal pH swab, and a stool sample at Day 14 and at Day 28. An additional vaginal swab sample will be collected at Day 35 to assess for probiotic strains persistence.

At the conclusion of the study, participants will be instructed to return any unused supplements to the study site.

ELIGIBILITY:
Inclusion criteria:

1. Be a healthy female between the ages of 18 and 40 years,
2. Have a regular and predictable menstrual cycle,
3. Be on an oral contraceptive,
4. Willing and able to consume a probiotic supplement for 4 weeks,
5. Willing and able to complete daily questionnaires online regarding dietary intake and general health and well-being, including gastrointestinal habits,
6. Willing to discontinue consumption of probiotics supplements and probiotic fortified products two weeks prior the beginning of the study and throughout the study,
7. Willing to discontinue consumption of fiber supplements,
8. Willing to provide a stool sample two times during the study,
9. Willing to provide one vaginal swab sample four times during the study,
10. Willing to provide one skin swab sample (skin between the vagina and the anus), three times during the study,
11. Typically have one stool per day,
12. Willing to complete a pregnancy test before consuming the study supplement.

Exclusion criteria:

1. Women who will be menstruating during the sample collection times,
2. Women who only use condoms, barrier, spermicide, or natural methods as their sole contraceptive method,
3. Women using any intrauterine device (IUD), birth control shot or implant,
4. Women who are lactating, know that they are pregnant, are attempting to get pregnant or test positive on a pregnancy test,
5. Pre-menopausal or menopausal women,
6. Women who have used any vaginal probiotics in the previous three months,
7. Use of oral or local antibiotics or antifungal within the past month,
8. Currently being treated for a severe chronic disease (cancer, renal failure, chronic inflammatory digestive or gastro-intestinal disease, immunodeficiency, etc.),
9. Women who have been diagnosed with any gynecological diseases or conditions (fibroma, endometriosis, etc.),
10. Women who have been diagnosed with secondary dysmenorrhea,
11. Women with intolerance, allergy or hypersensitivity to milk, soy or yeast,
12. With ongoing symptoms of vaginal and/or urinary tract infection,
13. Women using a treatment for vaginal sepsis or urosepsis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participant must menstruate regularly and consume an oral contraceptive.
Enrollment: 8 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

PRIMARY OUTCOMES:
Strains detection | Baseline, Day 14, Day 28, Day 35
  Change in presence or absence of the probiotic bacterial strains in the vaginal swab samples after 4 weeks of orally consuming the probiotic supplement.

SECONDARY OUTCOMES:
Strains viability | Baseline, Day 14, Day 28, Day 35
  Viability of the probiotic bacterial strains in the vaginal and skin swab samples.
Stool frequency | weekly, up to 6 weeks
  Average number of stools per week.
Stool consistency | weekly, up to 6 weeks
  Intestinal transit time as measured by the Bristol Stool Form Scale (BSFS). The BSFS is scored between 1 (hard stool) - 7 (liquid stool).
Stress | weekly, up to 6 weeks
  Measured daily on a scale between 1 (no stress) to 10 (extremely stressed).
Vaginal pH | Baseline, Day 14, Day 28
  Evolution of vaginal pH throughout intervention.
Strains detection in skin swabs | Baseline, Day 14, Day 28
  Presence or absence of the probiotic strains in the skin swab samples.
Strains persistence | Baseline, Day 35
  Presence or absence of the probiotic strains in the vaginal swab sample 1 week after the intervention has been completed.
Strains recovery in stool samples | Baseline, Day 28
  Change from baseline in the concentration of the probiotic strains in stool samples.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, Ph.D., Principal Investigator — University of Florida
Locations (1):
- Food Science and Human Nutrition Department and the Center for Nutritional Sciences, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No
After publications of the results, de-identified data will be shared with qualified researchers and scientists upon reasonable request to the sponsor including a detailed proposal of the intended use of the data, as per the Lallemand Health Solutions Inc. Policy on Clinical Trial Transparency and Data Sharing (available upon request).